CLINICAL TRIAL: NCT06228625
Title: Comparison of Rehabilitative Game Exercise and Body Awareness Therapy in Rotator Cuff Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ozlem Gorgulu Goksu, Physiotherapist,Master of Science (M.Sc.), Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMUogorgulugoksu1
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Syndrome
Keywords: Body Awareness; Body İmage; Exergame; Rotator cuff; Videogames

STUDY DESIGN:
Intervention Model Description: Randomize Controlled Double Blind Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Conventional exercise training will be given to the control group for 6 weeks, 5 days a week, for 45 minutes. Conventional exercises will be applied to this group under the supervision of a physiotherapist for 5 days in our unit.
  Interventions: Behavioral: Conventional Exercise Group
- Body Awareness Training Group (Experimental): After the first evaluation, the training group will be given basic body awareness exercise training for 6 weeks, 2 days a week, for 45 minutes. This group will be given to basic body awareness exercises under the supervision of a physiotherapist for 2 days in our unit. Individuals in this group will be applied basic body awareness exercisea program in addition to conventional exercises.
  Interventions: Behavioral: Body Awareness Training Group
- Rehabilitative Game Exercise Group (Experimental): Individuals in this group will be applied a video-based rehabilitative game exercise program in addition to conventional exercises. A digital game network called 'Active Arcade Game' will be used for rehabilitative game exercises. Rehabilitative Game Exercise Group for 6 weeks, 2 days a week, for 45 minutes. This group will be given to basic body awareness exercises under the supervision of a physiotherapist for 2 days in our unit.
  Interventions: Behavioral: Rehabilitative Game Exercise Group

INTERVENTIONS:
Behavioral: Conventional Exercise Group — * Wand Exercises (Shoulder flexion, abduction, extension, external, internal rotation *10 rep.)
  * Codmann Exercises (In each direction with front-back, right-left, clockwise and counterclockwise movements *10 rep.)
  * Finger Ladder (flexion and abduction directions * 10 rep.)
  * Strengthening Exercises (Shoulder flexion, abduction, extension, external, internal rotation *10 rep).
  * Posterior, anterior and inferior capsule stretching ,pectoral muscle stretching * 10 rep.
  Arms: Control Group
Behavioral: Body Awareness Training Group — * Supine: Body scan, contraction-relaxation exercises, strength recovery exercises combined with sound, stretching exercises, cross and star stretching.
  * Sitting: Teaching the correct body alignment while sitting, exercise to restore the correct body alignment,
  * Standing: Weight bearing exercises within stability limits, midline descent and elevation exercises, midline rotation exercises, wave motion, pushing movement combined with oblique weight bearing.
  Arms: Body Awareness Training Group
Behavioral: Rehabilitative Game Exercise Group — * Cone Knockout: The game requires touching the cones that appear alternately on the right and left within one minute.
  * Space Pong: It is required to play by hitting the ball with the right or left hand. It requires only upper extremity use and has seven abductions. Scoring is based on the ball hit.
  * Reaction: It is a game that requires touching the green dots that appear on the screen within a certain period. The points received vary depending on the speed of touching the dots. Points are lost when the red dots are touched.
  * Whack A Male: The player has 3 rights, and it requires using the upper extremity to hit the moles that come out of 5 holes at different times. A mole with a thorn on its head and a bomb should not be hit. Before the spiny mole emerges, a red light appears in the hole where it will emerge.
  Arms: Rehabilitative Game Exercise Group

SUMMARY:
Rotator cuff syndrome is one of the most common problems in the shoulder, starting as acute tendinopathy and progressing to partial and full thickness tears. Shoulder pain causes a decrease in shoulder joint movement, joint position sense, upper extremity function and quality of life. Among the most commonly used conservative treatment methods; Joint range of motion exercises, stretching exercises, strengthening exercises, mobilization and electrotherapy method are included.

Nowadays, with the widespread use of technology in rehabilitation, video-based games have begun to be used for rehabilitative purposes in addition to conservative approaches. Although the effectiveness of video-based games has been extensively studied in diseases such as cerebral palsy, stroke and parkinsonism, there are a limited number of studies in the field of orthopedic rehabilitation, especially in shoulder rehabilitation.

Basic body awareness therapy is used to treat chronic musculoskeletal-related painful conditions. In the literature, basic body awareness therapy has been studied in patient groups such as mental health, stroke patient groups, chronic musculoskeletal problems, chronic waist and neck pain, scoliosis and knee osteoarthritis. Studies have shown that the TBFT method provides improvements in individuals' body awareness, mobility in daily living activities, health-related quality of life, body image and pain intensity. However, no studies have been found in which basic body awareness therapy was used in the field of shoulder rehabilitation.

Our study aims to compare the effectiveness of a rehabilitative game exercise program and body awareness training in terms of pain, joint range of motion, shoulder functionality, proprioception, body awareness, shoulder-related quality of life, kinesiophobia and patient satisfaction in individuals with Rotator cuff syndrome.

DETAILED DESCRIPTION:
It is one of the most common problems in the shoulder, which begins as acute tendinopathy in rotator cuff surgery and can progress to partial and full thickness tears. The most commonly affected muscle is supraspinatus and infraspinatus, followed in second place.

The shoulder joint is an important and complex joint in terms of both mobility and stability. Having a wide joint range of motion makes stabilization of this joint difficult. Passive (bone, capsule, ligament) and active (muscles) structures play an important role in ensuring stability. The stabilization mechanism is under the control of the central nervous system. The sensorimotor system is responsible for all proprioceptive information, motor or neuromuscular responses and central integration, and plays a role in maintaining the balance of static and dynamic stabilizers around the joint.Proprioceptive sensory input is one of the most important structures of the sensorimotor system. Insufficiency in proprioceptive sense is one of the factors that predispose to injuries, and studies have shown that proprioceptive deficit is present in common pathologies of the shoulder such as shoulder instability, impingement syndrome, rotator cuff injuries, adhesive capsulitis and osteoarthritis. The first symptom that usually occurs in rotator cuff injuries is pain, and its incidence increases significantly with age.Shoulder pain and increasing shoulder joint movement limitation cause a decrease in shoulder active joint position sense (proprioception), upper extremity function and quality of life. Exercise prescription in general; It focuses on increasing the range of motion of the glenohumeral joint and the flexibility of the muscles in the region, providing scapular control and increasing the muscle strength of the shoulder area. Among the most commonly used conservative treatment methods; Joint range of motion exercises, stretching exercises, strengthening exercises, mobilization and electrotherapy method are included.

Today, with the widespread use of technology in rehabilitation, video-based games have begun to be used for rehabilitative purposes in addition to conservative approaches.

Products such as Nintendo Wii, Microsoft Kinect and Fizyosoft can be given as examples of video-based games. Video-based game exercise programs are defined as a combination of physical movements and games designed to increase the physical activity level and functionality of individuals. Although the effectiveness of video-based games in neurorehabilitation has been extensively studied in diseases such as cerebral palsy, stroke and parkinsonism, there are a limited number of studies in the field of orthopedic rehabilitation, especially in the treatment protocols of patients with rotator cuff injury and subacromial impingment syndrome.

Basic Body Awareness Therapy is an existential treatment approach targeting mind-body integrity that is frequently used in the rehabilitation of patients with psychiatric disorders and chronic musculoskeletal problems. Basic body awareness therapy is used in the treatment of painful conditions related to the chronic musculoskeletal system. In the literature, it has been seen that basic body awareness therapy has been studied in patient groups such as mental health, stroke patient groups, chronic musculoskeletal problems, chronic waist and neck pain, scoliosis and knee osteoarthritis. It has been shown in the studies examined that the basic body awareness therapy method, which provides integration of mind-body integrity, provides improvement in individuals' body awareness, mobility in daily living activities, health-related quality of life, body image and pain intensity findings. However, no studies have been found in which basic body awareness therapy was used in the field of shoulder rehabilitation.

The aim of our study is to compare the effectiveness of a rehabilitative game exercise program and body awareness training in terms of pain, joint range of motion, shoulder functionality, proprioception, body awareness, shoulder-related quality of life, kinesiophobia and patient satisfaction in individuals with Rotator cuff syndrome. In addition to conventional methods, the rehabilitative game exercise programWe predict that body awareness training will bring a different perspective to the field of shoulder rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial supraspinatus rupture by an Orthopedics and Traumatology specialist placement.
* Unilateral shoulder pain,
* Not having been involved in any physiotherapy program before due to shoulder problem,
* Body mass index (BMI) ≤ 30 kg/m²
* Cooperation of individuals

Exclusion Criteria:

* Having had previous shoulder surgery,
* Having received local corticosteroid injection/corticosteroid treatment in the last three months,
* Presence of a disease that will affect the neurological, cardiac, systemic, cognitive and visual systems,

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Pain Severity rated their feelings of pain on the line by themselves, thereby quantifying the pain.sual Analogue Scale | Baseline and after 6 weeks
  Participants pain intensities ranged from "0" (no pain) to "10" (unbearable pain) to 10 cm will be evaluated with the Visual Pain Scale. The pain intensity of the participants before and after the treatment was evaluated at rest and during activity.
Pain threshold | Baseline and after 6 weeks
  Algometer is a device used to evaluate the pain threshold, thanks to the pressure it applies. While increasing the pressure using the algometer, persons are asked to indicate at the first point where they feel pain or discomfort. The first point of discomfort is defined as the pain threshold of the individual.The first point of discomfort is defined as the individual's pain threshold point. When evaluating the pain thresholds of people participating in the study, their most sensitive areas will be taken as reference. Measurements will be repeated 3 times and their average will be taken.
Evaluation of joint range of motion | Baseline and after 6 weeks
  Baseline digital Absolute + Axis goniometer device will be used. Flexion, extension, abduction, internal and external rotation range of motion of the shoulder joint will be evaluated in degrees. For each joint range of motion value, 3 consecutive measurements will be taken and the average value will be recorded.
Evaluation of Joint Position Sense | Baseline and after 6 weeks
  Active angle repetition test for shoulder joint position sense will be performed with the smartphone goniometer application. 40° and 100° elevation angles will be used in the scapular plan, which are frequently preferred in the literature. For the evaluation, first of all, the participants will be asked to passively perform a 40° elevation movement on one shoulder in the scapular plane while their eyes are open and they will be asked to learn this angle. Then, the participants will raise their shoulders to 40° elevation 3 more times with their eyes closed, wait 10 seconds to teach this angle, and then return to the starting position.The test will be repeated 6 times and individuals will rest for 5 seconds between each repetition. All applications were repeated for a shoulder elevation angle of 100°. The test was performed at 40° and 100° shoulder elevation on both shoulders.

SECONDARY OUTCOMES:
Rotator Cuff Quality of Life | Baseline and after 6 weeks
  It is a questionnaire that evaluates the quality of life in rotator cuff injuries. It is a disease-specific questionnaire and is distinctive in assessing quality of life. It is a questionnaire consisting of 34 questions and 5 subparameters that evaluates the physical symptoms of the disease, work activities, daily living activities, social and emotional status. Each question is calculated out of 100 points and the total score is expressed as a percentage.
American Shoulder and Elbow Surgeons (ASES) | Baseline and after 6 weeks
  American Shoulder and Elbow Surgeons (ASES) created the ASES questionnaire in order to develop a standardized method for evaluating shoulder function. The goal was to design a questionnaire that was easy to use, assessed function, and was entirely based on patient self-evaluation. The ASES score totals 100 points and allocates 50 points for measuring function and 50 points for pain.
Body Awareness Questionnaire | Baseline and after 6 weeks
  The body awareness questionnaire is a 18 item scale, with the total scale score calculated as a sum of the items. Items are scored on a 1-7 scale, with the total scale score calculated as a sum of the items. The questions with asterisks are reverse scored. This means that for example, if someone scored 1 it would now be a score of 5.
Body Image Survey (BIA) | Baseline and after 6 weeks
  BIA was used to measure the patients' level of satisfaction with their body image. BIA consists of a person's body parts or functions.It is a scale that determines satisfaction. It was shown in the study by Hovardaoğlu et al. that the scale is valid and reliable in Turkish.
The Tampa Scale for Kinesiophobia (TSK) | Baseline and after 6 weeks
  The Tampa Scale for Kinesiophobia (TSK) is a self-report questionnaire that is used to assess an individual's fear of movement or re-injury. The TSK consists of 17 items that ask respondents to rate their level of agreement with statements related to the fear of movement or re-injury. A high score from the scale indicates a high level of kinesiophobia.
Patient Satisfaction Evaluation | After 6 weeks
  How much of the applied treatment meets the patients' expectations can be simply asked by asking "what is the percentage of your recovery rate with the applied treatment?" and "What is the percentage of the treatment applied that meets your expectations?" It was evaluated with two questions. Participants' answers were recorded as percentage values.

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem Görgülü Göksu, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No